CLINICAL TRIAL: NCT02189824
Title: Chemotherapy Followed by Infusion of Partially HLA Matched Unrelated Donor Cells for Patients With AML Who Are Ineligible for Stem Cell Transplantation
Acronym: SCRAMBLE
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sydney (Other)
Collaborators: Melbourne Health (Other); Royal Brisbane and Women's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCTL141501; PG1061252 (Other Grant/Funding Number: Australian NHMRC)
Record Dates: First submitted 2014-07-11; First posted 2014-07-15 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Acute Myeloid Leukaemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Infusion of partially matched unrelated donor cells (Experimental)
  Interventions: Biological: Partially HLA-matched unrelated donor cells

INTERVENTIONS:
Biological: Partially HLA-matched unrelated donor cells

SUMMARY:
A phase 1 study of infusion of partially HLA matched unrelated donor blood or marrow cells (microtransplantation) following consolidation chemotherapy in patients with AML that are not suitable for allogenic stem cell transplantation.

DETAILED DESCRIPTION:
To determine the safety and tolerability of co-administration of partially HLA antigen matched unrelated donor cryopreserved donor lymphocytes (microtransplantation) with chemotherapy for patients with high risk acute myeloid leukaemia ineligible or unsuitable for high dose chemotherapy and stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed AML not considered suitable for allogenic stem cell transplant on the basis of age or co-morbidities
2. Complete morphological remission following 1-2 cycles of induction chemotherapy consisting of an anthracycline/cytosine arabinoside combination
3. Availability of cryopreserved donor stem cells or bone marrow with appropriate HLA matching
4. Adequate hepatic and renal function
5. Estimated life expectancy of at least 6 months
6. Patient has given informed consent or in the event of a patient not able to give informed consent, consent has been given according to hospital procedures in force at the time of trial

Exclusion Criteria:

1. Patient not in morphological remission following 2 cycles of induction chemotherapy
2. Use of fludarabine or other purine analogue during remission induction or use of any major immunosuppressive medication or any other immunomodulatory agent including thalidomide, lenalidomide, or azacitidine immediately prior to concurrent with administration of chemotherapy for AML or during or in the 3 months after administration of partially HLA matched 3rd party cells
3. Absence of a cryopreserved donor stem cell or bone marrow product with appropriate matching
4. Presence of significant hepatic, renal or other major organ dysfunction
5. Uncontrolled infection or bleeding prior to commencement of consolidation chemotherapy
6. Privately insured in or outpatient on the day the consent is signed and the days that cryopreserved partially HLA matched donor cells are infused

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute graft versus host disease within 60 days of completion of final infusion of donor lymphocytes | 60 days

SECONDARY OUTCOMES:
Duration of post chemotherapy cytopenias | 60 days
Remission rate | 12 months
Duration of complete remission | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Westmead Hospital Department of Haematology, Westmead, Sydney, New South Wales, Australia